CLINICAL TRIAL: NCT05346471
Title: Infra- and Supratentorial Neuromonitoring in Patients With Posterior Fossa Lesions: DUAL-ICP Trial
Brief Title: Infra- and Supratentorial Neuromonitoring
Acronym: DUAL-ICP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCH -11112018
Record Dates: First submitted 2022-03-30; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-01

CONDITIONS: Intracranial Pressure Increase; Posterior Fossa Lesion; Posterior Fossa Hemorrhage
Keywords: Infratentorial Neuromonitoring
MeSH Terms: conditions — Intracranial Hypertension; Intracranial Hemorrhages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute posterior fossa lesions (Other): Subjects will receive additional multimodal infratentorial neuromonitoring
  Interventions: Device: Multimodal neuromonitoring

INTERVENTIONS:
Device: Multimodal neuromonitoring — Multimodal neuromonitoring accounts for intraparenchymatous ICP probe, brain tissue oxygen probe and/or cerebral microdialysis device

SUMMARY:
Invasive neuromonitoring of intracranial pressure (ICP) is an important element of neurosurgical critical care that is used primarily as an indicator of adequate cerebral perfusion in patients, when clinical observation is not an option. Due to the constraint in size and the critical structures within the posterior fossa, detection of intracranial pressure particularly in the postoperative phase has been deemed desirable in patients with surgery in this region, particularly in those subjected to prolonged procedures and critical care.

The posterior fossa is an anatomically constricted compartment with narrow spaces and intracranial hypertension quickly leads to brainstem damage and neurological dysfunction. ICP in the supratentorial space not necessarily correlates with ICP in the infratentorial space. Some authors claim that it would be beneficial to measure ICP in infratentorial space after posterior fossa surgery in some cases.

The relationship between the intracranial pressure profiles in the supratentorial and infratentorial compartments remain unclear. After a neurosurgical operation in the posterior fossa there are most likely pressure differences between supra- and infratentorial spaces. It is well known that the pressure within the skull is unevenly distributed, with appreciable ICP gradients.

Thus, the investigators intend to apply the intracranial multimodal monitoring in both infratentorial and supratentorial compartments simultaneously. Such coincident measurements most likely will be the most sensitive way to assess focal swelling, ischemia and tissue perfusion, or other relevant complications in the posterior fossa structures.

The goal of this study is to test whether direct infratentorial monitoring is a more efficacious method for detecting dynamic changes in the operative compartment and whether it is safe, in view of the critical structures within the region.

DETAILED DESCRIPTION:
Invasive neuromonitoring of intracranial pressure (ICP) is an important element of neurosurgical critical care that is used primarily as an indicator of adequate cerebral perfusion in patients, when clinical observation is not an option. Due to the constraint in size and the critical structures within the posterior fossa, continuous detection of postoperative pressures has been deemed desirable in patients with surgery in this region, particularly in those subjected to prolonged procedures and critical care.

The posterior fossa is an anatomically constricted compartment with narrow spaces and intracranial hypertension quickly leads to brainstem damage and neurological dysfunction. ICP in the supratentorial space not necessarily correlates with ICP in the infratentorial space. Some authors claim that it would be beneficial to measure ICP in infratentorial space after posterior fossa surgery in some cases.

In patients whose neurological examination results may be inconclusive or limited, it is valuable to have a reliable alternative method of evaluation. It is generally accepted that continuous ICP monitoring is very important to determine the timing of surgery and to prevent secondary brain damage caused by increased ICP.

There have been few clinical studies in which simultaneous pressures were recorded above and below the tentorium in patients with intracranial pathology. Yet, the relevance of infratentorial neuromonitoring remains largely unclear. So far, the placement of ICP probes in the posterior fossa seems to carry very low morbidity. Furthermore, to rely on autonomic changes, neurological deterioration, or measurements of only the supratentorial compartment as a sign of relevant complications in the posterior fossa highly narrows the temporal margin of safety for the institution of treatment. Comprehensive evaluation of possible risks of posterior fossa lesions and their treatments is crucial. Of note, immediate detection of treatment-related complications is often challenging, still being able to avoid permanent neurological sequelae. The application of the advanced neuromonitoring in the posterior fossa may be supportive in achieving this difficult goal and may provide objective assessments of procedure-related complications.

Therefore, the data generated by our prospective trial can be expected to be beneficial in individualized treatment plans. It is a relatively novel approach to intracranial multimodal neuromonitoring. The application of infratentorial probes offers potential for better understanding of lesion maturation and progression, clinical deterioration, and monitoring the effect of treatments.

The investigators hypothesize that additional multimodal infratentorial neuromonitoring will be of high clinical value detecting any relevant complication and giving detailed insight in pathophysiological interactions in posterior fossa lesions.

ELIGIBILITY:
Inclusion Criteria:

* Posterior fossa lesions with anticipated prolonged neurointensive critical care
* Patients older than 18 years
* Informed consent if applicable (unconscious patients will be also enrolled)
* No existing exclusion criteria

Exclusion Criteria:

* Coagulation disorders
* Age < 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of device-related events [Safety and Tolerability] | From implementation until removing of infratentorial multimodal neuromonitoring, assessed up to 30 days
  All device-related events (infections, tissue irritation, haemorrhage along device trajectory, dural leaks etc.) will be noted and reported, even if no clinical consequence will ensue
Correlation | As long as neuromonitoring is indicated, assessed up to 30 days
  Correlation analysis of supra- and infratentorial measures
Glasgow Outcome Scale (GOS) after 3 months | Assessed 3 months after initial treatment
  GOS to asses the potential influence of infratentorial monitoring measures on clinical outcome (GOS 1-3 poor outcome; GOS 4-5 good outcome)
Glasgow Outcome Scale (GOS) after 6 months | Assessed 6 months after initial treatment
  GOS to asses the potential influence of infratentorial monitoring measures on clinical outcome (GOS 1-3 poor outcome; GOS 4-5 good outcome)
Glasgow Outcome Scale (GOS) after 9 months | Assessed 9 months after initial treatment
  GOS to asses the potential influence of infratentorial monitoring measures on clinical outcome (GOS 1-3 poor outcome; GOS 4-5 good outcome)
modified Ranking Scale (mRS) after 3 months | Assessed 3 months after initial treatment
  mRS as alternative outcome measure to asses the potential influence of infratentorial monitoring measures on clinical outcome (mRS 0-6; the higher the worse the outcome)
modified Ranking Scale (mRS) after 6 months | Assessed 6 months after initial treatment
  mRS as alternative outcome measure to asses the potential influence of infratentorial monitoring measures on clinical outcome (mRS 0-6; the higher the worse the outcome)
modified Ranking Scale (mRS) after 9 months | Assessed 9 months after initial treatment
  mRS as alternative outcome measure to asses the potential influence of infratentorial monitoring measures on clinical outcome (mRS 0-6; the higher the worse the outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ondra Petr, MD PhD, Principal Investigator — Consultant - Faculty/Staff
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No
Collection of data and publish results

REFERENCES:
- [Background] Slavin KV, Misra M. Infratentorial intracranial pressure monitoring in neurosurgical intensive care unit. Neurol Res. 2003 Dec;25(8):880-4. doi: 10.1179/016164103771954014. PMID 14669535
- [Background] Khan A, Borg N, Shenouda E. Posterior fossa ICP monitoring: a tale of two compartments. Br J Neurosurg. 2021 Apr;35(2):129-132. doi: 10.1080/02688697.2020.1765974. Epub 2020 May 15. PMID 32410470
- [Background] Rosenwasser RH, Kleiner LI, Krzeminski JP, Buchheit WA. Intracranial pressure monitoring in the posterior fossa: a preliminary report. J Neurosurg. 1989 Oct;71(4):503-5. doi: 10.3171/jns.1989.71.4.0503. PMID 2795169
- [Background] Moyse E, Ros M, Marhar F, Swider P, Schmidt EA. Characterisation of Supra- and Infratentorial ICP Profiles. Acta Neurochir Suppl. 2016;122:37-40. doi: 10.1007/978-3-319-22533-3_7. PMID 27165873
- [Background] LANGFITT TW, WEINSTEIN JD, KASSELL NF, SIMEONE FA. TRANSMISSION OF INCREASED INTRACRANIAL PRESSURE. I. WITHIN THE CRANIOSPINAL AXIS. J Neurosurg. 1964 Nov;21:989-97. doi: 10.3171/jns.1964.21.11.0989. No abstract available. PMID 14238966
- [Background] Wolfla CE, Luerssen TG, Bowman RM, Putty TK. Brain tissue pressure gradients created by expanding frontal epidural mass lesion. J Neurosurg. 1996 Apr;84(4):642-7. doi: 10.3171/jns.1996.84.4.0642. PMID 8613857
- [Background] Vanaclocha V, Saiz-Sapena N, Rivera-Paz M, Herrera JM, Ortiz-Criado JM, Verdu-Lopez F, Vanaclocha L. Can we safely monitor posterior fossa intracranial pressure? A cadaveric study. Br J Neurosurg. 2017 Oct;31(5):557-563. doi: 10.1080/02688697.2017.1332336. Epub 2017 May 25. PMID 28539078
- [Background] Rosner MJ, Becker DP. ICP monitoring: complications and associated factors. Clin Neurosurg. 1976;23:494-519. doi: 10.1093/neurosurgery/23.cn_suppl_1.494. PMID 975699
- [Background] Maas AI, Schouten JW, Stocchetti N, Bullock R, Ghajar J. Questioning the value of intracranial pressure (ICP) monitoring in patients with brain injuries. J Trauma. 2008 Oct;65(4):966-7. doi: 10.1097/TA.0b013e318184ee7b. No abstract available. PMID 18849824
- [Background] Saul TG, Ducker TB. Effect of intracranial pressure monitoring and aggressive treatment on mortality in severe head injury. J Neurosurg. 1982 Apr;56(4):498-503. doi: 10.3171/jns.1982.56.4.0498. PMID 6801218
- [Background] Piek J, Bock WJ. Continuous monitoring of cerebral tissue pressure in neurosurgical practice--experiences with 100 patients. Intensive Care Med. 1990;16(3):184-8. doi: 10.1007/BF01724800. PMID 2351779
- [Derived] Petr O, Ho WM, Petutschnigg T, Krigers A, Treichl SA, Preuss-Hernandez C, Brawanski K, Helbok R, Thome C. Link between both infratentorial and supratentorial intracranial pressure burdens and final outcome in patients with infratentorial brain injury. J Neurosurg. 2023 Apr 28;139(5):1430-1438. doi: 10.3171/2023.1.JNS221806. Print 2023 Nov 1. PMID 37119097

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT05346471/Prot_SAP_000.pdf